CLINICAL TRIAL: NCT07106307
Title: Evaluation of the Effect of Different Root Canal Obturation Techniques on the Success of Root Canal Treatment in Teeth With Apical Periodontitis
Brief Title: Evaluation of Different Root Canal Obturation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ASLI USTA TAHMAZ, Principal Investigator, Department of Endodontics, Medipol University, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6496
Record Dates: First submitted 2025-07-12; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Apical Periodontitis; Periapical Lesion
Keywords: Apical Periodontitis; Periapical Healing; Bioseramic sealer; Epoxy Resin Based Sealer; Warm Vertical Compaction
MeSH Terms: conditions — Periapical Periodontitis | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold lateral compaction with AH Plus (Epoxy Resin Based Sealer) (Experimental): Root canal obturation will be performed using the cold lateral compaction technique with AH Plus epoxy-resin based sealer.
  Interventions: Other: Epoxy Resin-Based Sealer; Procedure: Cold Lateral Compaction
- Cold lateral compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer) (Experimental): Root canal obturation will be performed using the cold lateral compaction technique with AH Plus Bioceramic sealer.
  Interventions: Other: Bioceramic Sealer; Procedure: Cold Lateral Compaction
- Warm vertical compaction with AH Plus (Epoxy Resin Based Sealer) (Experimental): Root canal obturation will be performed using the warm vertical compaction technique with AH Plus epoxy-resin based sealer.
  Interventions: Procedure: Warm Vertical Compaction; Other: Epoxy Resin-Based Sealer
- Warm vertical compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer) (Experimental): Root canal obturation will be performed using the warm vertical compaction technique with AH Plus Bioceramic sealer.
  Interventions: Other: Bioceramic Sealer; Procedure: Warm Vertical Compaction

INTERVENTIONS:
Other: Bioceramic Sealer — This intervention involves the use of Bioceramic Sealer during root canal obturation. The sealer will be combined with the cold lateral compaction or warm vertical compaction technique depending on the study arm.
  Arms: Cold lateral compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer); Warm vertical compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer)
Procedure: Warm Vertical Compaction — Warm vertical obturation is performed using a heat delivery device, which thermosoftens gutta-percha and allows vertical compaction into the root canal system. This technique will be used in combination with either resin-based or bioceramic sealers, depending on the study group.
  Arms: Warm vertical compaction with AH Plus (Epoxy Resin Based Sealer); Warm vertical compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer)
Other: Epoxy Resin-Based Sealer — This intervention involves the use of an epoxy resin-based root canal sealer during root canal obturation. The material will be applied in combination with either cold lateral compaction or warm vertical compaction techniques, depending on the study group.
  Arms: Cold lateral compaction with AH Plus (Epoxy Resin Based Sealer); Warm vertical compaction with AH Plus (Epoxy Resin Based Sealer)
Procedure: Cold Lateral Compaction — Cold lateral compaction is a root canal obturation technique in which a master gutta-percha cone is placed to working length and compacted laterally using a finger spreader. This method will be used in combination with either resin-based or bioceramic sealers, depending on the study group.
  Arms: Cold lateral compaction with AH Plus (Epoxy Resin Based Sealer); Cold lateral compaction with AH Plus Bioceramic (Calcium Silicate Based Sealer)

SUMMARY:
The aim of this clinical study is to evaluate the effect of root canal filling, which is the last stage of root canal treatment (RCT), on the post-operative pain level on single rooted permanent teeth with wide lesions with apical periodontitis, and the effect on the healing of the periapical tissue and lesion by comparing periapical radyography images, which was taken at the beginning and after one year.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of different root canal filling techniques on postoperative pain levels and the healing of periapical tissues in teeth with periapical lesions, using periapical radiographic imaging. Specifically, the effects of resin-based sealers, bioceramic-based sealers, and two obturation techniques-cold lateral compaction and warm vertical compaction-will be compared. Postoperative pain will be assessed using VAS (Visual Analog Scale) and VRS (Verbal Rating Scale) following the final stage of root canal treatment in incisor and premolar teeth with single roots. Additionally, the healing of periapical lesions will be evaluated by comparing periapical radiographs taken at baseline and at a one-year follow-up. To date, no study has been found in the literature that evaluates these specific combinations of materials and techniques using periapical radiographic imaging.

The study includes four experimental groups based on the combination of obturation technique and sealer type as follows:

Group 1: Cold lateral compaction with AH Plus (epoxy resin-based sealer)

Group 2: Cold lateral compaction with AH Plus Bioceramic (calcium silicate-based sealer)

Group 3: Warm vertical compaction with AH Plus

Group 4: Warm vertical compaction with AH Plus Bioceramic

All treatments will be performed under standardized clinical conditions by an experienced endodontist using a rubber dam in aseptic conditions. Chemomechanical preparation will be done using rotary NiTi instruments and an irrigant protocol consisting of Sodium Hypochlorite (NaOCl), Ethylenediaminetetraacetic Acid (EDTA), and distilled water using Ultrasonic irrigation device. Root canal filling will be performed in a single visit for all patients.

VAS and VRS scores will be recorded at multiple time points postoperatively: immediately after treatment, and at 6, 12, 18, 24, 48, and 72 hours, as well as at 1 week and 1 month. Pain diaries will be provided to all participants.

Radiographic evaluation will be performed using standardized periapical radiographs taken with a parallel technique. Periapical healing will be assessed by comparing lesion size at baseline and at 1 year by two blinded observers.

This study aims to provide clinical data that may guide endodontic decision-making regarding the choice of sealer and obturation technique, particularly in teeth with pre-existing periapical pathology.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted anterior and premolar teeth with radiographically confirmed periapical lesions classified as Periapical Index (PAI) scores of 4 or 5 will be included in the analysis
* Age between 18 and 60 years
* Systemically healthy individuals
* To be able to read and sign the informed consent form
* Physical and mental fitness to undergo treatment
* Willingness to attend all follow-up sessions

Exclusion Criteria:

* Patients with systemic diseases classified as ASA III or higher
* Presence of severe periodontal disease (probing depth >4 mm)
* Use of analgesics within the last 12 hours or antibiotics within the past month before the treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Periapical Healing | From end of treatment to 1 year
  The primary outcome of this study is periapical healing. It will be assessed radiographically using standardized periapical images (taken with the parallel technique), captured preoperatively and at the 1-year follow-up, and evaluated using the Periapical Index (PAI) score by two blinded observers. The PAI score ranges from 1 (healthy periapical structures) to 5 (severe periodontitis).

SECONDARY OUTCOMES:
Post Operative Pain İntensity | From end of treatment to 6, 12, 18, 24, 48, and 72 hours; 7 days; and 1 month after root canal treatment
  The secondary outcome is postoperative pain intensity. Pain will be assessed at multiple time points (6, 12, 18, 24, 48, and 72 hours, and at 1 week and 1 month post-treatment) using Visual Analog Scale (VAS) where 0 represents "no pain" and 10 represents "worst imaginable pain".
Post Operative Pain Intensity | From end of treatment to 6, 12, 18, 24, 48, and 72 hours; 7 days; and 1 month after root canal treatment
  The secondary outcome is postoperative pain intensity. Pain will be assessed at multiple time points (6, 12, 18, 24, 48, and 72 hours, and at 1 week and 1 month post-treatment) using Verbal Rating Scale (VRS), which categorizes pain into four levels: 0 (no pain), 1 (mild), 2 (moderate), and 3 (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), including all IPD that underlie the results reported in the publication
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared starting 6 months after publication.
Access Criteria: Qualified researchers may request access to all de-identified individual participant data (IPD) and study protocols. Access will be granted upon reasonable request by contacting the corresponding author via email and after signing a data sharing agreement